CLINICAL TRIAL: NCT00447889
Title: A Clinical Study of Gadoteric Acid in Non-Coronary Magnetic Resonance (MR)
Brief Title: A Clinical Study of Gadoteric Acid in Non-Coronary Magnetic Resonance (MR) Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: DGD-44-042
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Arterial Occlusive Disease
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gadoteric acid

SUMMARY:
This is a clinical study of gadoteric acid in non-coronary MR angiography.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least the age of legal maturity
* Strongly suspected of having non-coronary arterial disease, detected clinically
* Scheduled to undergo x-ray angiography examination
* Female patients must be using effective contraception or be surgically sterilized or post-menopausal.
* Females of childbearing potential must have a documented negative urine pregnancy test.

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI)
* Any metallic medical device in the vascular territory for which the patient is to undergo imaging examinations
* Congenital morphologic vascular abnormalities
* Known allergy to gadolinium chelates
* Pregnant, breast feeding, or planning to become pregnant during the trial
* Received a gadolinium complex within 2 days or iron oxide nanoparticles within 7 days before the gadoteric acid-enhanced magnetic resonance angiography (MRA) examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Dubourdieu, PhD, Study Chair — Guerbet
Locations (1):
- Asan Medical Center, Seoul, South Korea